CLINICAL TRIAL: NCT05318560
Title: Comparison of the Efficacy of Local Anesthetic and Ozone Injection in Patients With Myofascial Pain Syndrome
Brief Title: Efficacy of Local Anesthetic and Ozone Injection in Patients With Myofascial Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Hakan Alkan, Clinical Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PamukkaleU-Simsek-003
Record Dates: First submitted 2022-03-30; First posted 2022-04-08 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Myofascial Pain Syndrome; Ozone
Keywords: Ozone; Pain
MeSH Terms: conditions — Myofascial Pain Syndromes; Pain | interventions — Lidocaine; Ozone; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Local anesthetic injection (Active Comparator): Patients will be injected with lidocaine and given upper trapezius muscle stretching exercises. Lidocaine injection 2cc 2% will be administered to all patients using a 26 gauge, 0.45x13 mm disposable sterile needle to the affected trigger point.
  Interventions: Drug: Lidocaine 2% Injectable Solution; Other: stretching exercise
- Ozone injection (Active Comparator): Ozone injection will be performed on patients and upper trapezius muscle stretching exercises will be given. 8 cc of oxygen/ozone gas at a concentration of 15 µg/mL will be injected into the trigger point.
  Interventions: Drug: Ozone; Other: stretching exercise
- Stretching exercise (Active Comparator): Patients will be given a home program that includes upper trapezius muscle stretching exercises. Upper trapezius stretching exercises will be performed twice a day for at least 15 seconds, ten sets each time, for three weeks, with one hand on the patient's back and the other hand holding the side of the head and tilting it to the side until a slight tension is felt. The exercises will be explained in the text, visual and verbal forms with the exercise form.
  Interventions: Other: stretching exercise

INTERVENTIONS:
Drug: Lidocaine 2% Injectable Solution — for MPS
  Other Names: jetokain simplex
  Arms: Local anesthetic injection
Drug: Ozone — for MPS
  Arms: Ozone injection
Other: stretching exercise — for MPS

SUMMARY:
In this study, the investigators planned to compare local anesthetic injection added to stretching exercise, ozone injection treatment added to stretching exercise, and only stretching exercise in patients with upper trapezius muscle myofascial pain syndrome.

DETAILED DESCRIPTION:
The investigators will recruit 72 patients with at least one trigger point in the upper trapezius muscles and a clinically confirmed diagnosis of myofascial pain syndrome (MAS) (according to Travell-Simons' criteria) admitted to the physical medicine and rehabilitation outpatient clinic.

Age, gender, occupation, medications, duration of diagnosis, body mass index, comorbidity, functional status and pain of these patients will be questioned. Patients will be randomly divided into three groups. A total of 3 consecutive weeks of treatment were planned.

ELIGIBILITY:
Inclusion Criteria:

* With at least one trigger point in the upper trapezius muscles and a clinically confirmed diagnosis of MPS

Exclusion Criteria:

* Presence of any cervical radiculopathy or a history of degenerative conditions
* Presence of any cervical surgery or trauma in the past year,
* History of injection for the treatment of MAS in the last 6 months,
* Cognitive disorder,
* Rheumatological disease, fibromyalgia,
* History of metabolic diseases such as hypothyroidism and diabetes mellitus

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2022-09-10 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Change from baseline VAS at the 1st week after the treatment.
  The pain score will be measured using a 10 cm millimetric visual analog scale (VAS), where patients are asked to mark the degree of pain intensity from 0 (no pain) to 10 (worst pain imaginable) before and after treatment.

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | Change from baseline VAS at the 1st week after the treatment.
  NDI was assessed by the neck pain questionnaire that included 10 questions regarding the severity of neck pain, its impact on sleeping, driving, etc. Each question was scored from 0 to 5 and the total score was measured from 50 and was finally reported in percent (%). A higher percentage of NDI was an indicator of more disability and pain.
Range of motion (ROM) | Change from baseline VAS at the 1st week after the treatment.
  Range of motion (ROM) in neck lateral flexion movement measured according to the maximum angle that the patient could laterally bend his or her neck to the right and left side, using three consecutive times of goniometry and recording maximum value of them. Mean of the highest values of both directions was recorded as the final amount.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Alkan, Prof., Study Director — Pamukkale University